CLINICAL TRIAL: NCT07111026
Title: Sisters of Heart (Hermanas de Corazón): A Community Health Worker Initiative for Improving Heart Health in Migrant Farmworker Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Erin Ferranti, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00008487; 1R01NR021664-01 (NIH)
Record Dates: First submitted 2025-07-22; First posted 2025-08-08 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Occupational Stress; Gender Related Stress; Social Isolation; Hypertension; Pre Diabetes; Diabetes; Obesity
Keywords: occupational stress; gender related stress; social isolation; psychological stress; cardiometabolic health; social determinants of health
MeSH Terms: conditions — Occupational Stress; Social Isolation; Hypertension; Glucose Intolerance; Diabetes Mellitus; Obesity; Stress, Psychological

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sisters of Heart (Experimental)
  Interventions: Behavioral: Sisters of Heart
- Basic group (Other): Participants randomized to the Basic Intervention will have the option of crossing over to Sisters of Heart (Hermanas de Corazón's) intervention after their 3-month data collection is completed
  Interventions: Behavioral: Basic intervention

INTERVENTIONS:
Behavioral: Sisters of Heart — The intervention consists of ten weekly, 60-75-minute in-person peer support group sessions led by trained community health workers/promotoras (CHWs/Ps), with 6-10 participants per group. Sessions will be semi-structured, covering AHA Life's Essential 8 (LE8), stress management, and individualized topics based on participant priorities and social needs identified through surveys or group discussions. Each session includes stress management, core educational content, and time for addressing participant-driven issues. CHWs/Ps will also provide individualized support outside the sessions through direct community resource navigation, including phone or in-person "warm handoffs" to needed services.
  Other Names: Hermanas de Corazon
  Arms: Sisters of Heart
Behavioral: Basic intervention — The Basic intervention will include assessment of AHA LE8, provision to participants of results of 1) their baseline AHA LE8 assessments, including lab results, 2) written/online information with pertinent AHA LE8 health education content, 3) stress management educational materials, and 4) written information about the Ellenton Migrant Farm Worker Clinic and a community resource list
  Arms: Basic group

SUMMARY:
The goal of this hybrid Type 1 effectiveness-implementation trial is to test the extent to which a peer support and community resource navigation intervention improves psychological well-being, addresses social determinants of health and thus reduces cardiometabolic risk among rural, migrant, low-income farmworker women aged 18-45 years. The main questions it aims to answer are:

* If and to what extent does the intervention reduce stress, social isolation, and psychological distress by improving social support and access to needed resources?
* If and to what extent does the intervention improve cardiometabolic health, measured by the American Heart Association's Life's Essential 8 (LE8) score?

Researchers will compare the CHW-led Sisters of Heart (Hermanas de Corazón) intervention to a Basic intervention (LE8 assessment and resource information) to assess the effect of peer support and community resource navigation on heart health outcomes.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death in U.S. women, with a concerning rise in CVD mortality among women under 65-particularly those aged 35-44. Rural, migrant farmworker women face disproportionate risk factors and health disparities related to CVD, yet they remain underrecognized and underserved in prevention efforts. Only 44% of women recognize CVD as their top health threat. Although just 6% of Latinas have been diagnosed with CVD, they experience higher rates of obesity (48% vs. 38%) and type 2 diabetes (13% vs. 6%) compared to non-Latina White women.

Women farmworkers in rural areas face a compounded risk due to the convergence of biological, social, and structural factors. They are more likely to enter pregnancy with suboptimal cardiometabolic health and are at greater risk of gestational complications like preeclampsia and gestational diabetes, both of which significantly elevate future CVD risk. Cardiometabolic risks in the preconception and perinatal periods are strong predictors of both maternal mortality and lifelong CVD.

Improving cardiovascular health (CVH) in reproductive-age women is crucial to reducing maternal morbidity and long-term CVD burden. Many women's CVD risks go undiagnosed until pregnancy, underscoring the need for earlier prevention. The American Heart Association's Life's Essential 8 (LE8) provides a validated framework to measure and improve CVH. Yet, data show that only 1 in 5 U.S. Hispanic adults has high CVH, with Hispanic women scoring lower on diet, physical activity, and BMI metrics.

To address this, the study proposes a Community Health Worker (CHW)-led peer support intervention, Sisters of Heart (Hermanas de Corazón), targeting rural, low-income, reproductive-aged women farmworkers. While peer support interventions have demonstrated success in predominantly White, middle-aged populations and other health domains among underserved groups (e.g., cancer screening, postpartum wellness), no tailored CVD peer-support model currently exists for this high-risk population.

The Type 1 Hybrid Effectiveness-Implementation Design is ideally suited to this work. It allows for rigorous testing of the intervention's impact on CVH while simultaneously identifying barriers and facilitators to real-world implementation in rural farmworker settings. The study will fill an urgent gap by:

* Tailoring a culturally and linguistically appropriate intervention to Latina farmworkers
* Embedding trauma-informed care into CVD prevention
* Addressing SDOH-related stress and unmet needs
* Empowering CHWs to support peer behavior change and health system navigation
* Laying the groundwork for scaling and sustaining community-based CVH strategies in an underserved setting

ELIGIBILITY:
Inclusion Criteria:

* self-identified female employed as a migrant farmworker;
* Fluent in Spanish or English verbal literacy
* Planning to be in the geographic area for a minimum of 6 months.

Exclusion Criteria:

* Cognitive or psychological impairment precluding informed consent and/or active participation in the study due to substance use, neurologic, or other disorder
* Pregnant or breastfeeding.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 250 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in cardiometabolic health | T-0 (Baseline) ,T2 (3 months), T3 (6 months), T4 (7-9 months)
  The AHA's Life's Essential 8 score will be used to assess cardiometabolic health. The 8 components include 4 health behaviors (self-report) and 4 health factors (objective data).
  Each component is assigned 0-100 points per AHA LE8 scoring instructions. The total score is calculated as the mean of the 8 scores; higher total LE8 scores indicate greater adherence to health-promoting behaviors and factors.
Change in diet | Baseline, End of study (3 months)
  Diet will be assessed with the 23-item Mediterranean Eating Pattern for Americans (MEPA) III Questionnaire, adapted from the Mediterranean Diet Adherence Scale. MEPA assesses accordance with the Mediterranean-like diet pattern and asks about consumption of vegetables, nuts and seeds, fruits, fats and oils, meat and fish, dairy, beans and grains, desserts and fast food, and beverages
  Higher scores reflect greater adherence.
Change in physical activity | Baseline, End of study (3 months)
  Physical activity will be assessed with the 27-item International Physical Activity Questionnaire (IPAQ), a seven-day physical activity recall used in several large-scale studies and validated for use with Spanish-speaking communities in the US. A composite measure of physical activity will be derived based on the number of moderate to vigorous physical activity [5-8 metabolic equivalents (METs)] events the participant had in a typical week
Change in nicotine consumption | Baseline, End of study (3 months)
  Nicotine will be assessed in the health history survey. Questions include the history of current or ever smoked, the number of cigarettes smoked per day, and whether they live with an active smoker
Change in Sleep | Baseline, End of study (3 months)
  Sleep will be assessed with the Pittsburgh Sleep Quality Index (PSQI), a validated scale consisting of 7 components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medications, and daytime dysfunction.
  Each component is scored from 0 to 3, with higher scores indicating poorer sleep quality. The global PSQI score ranges from 0 to 21, and a score greater than 5 typically indicates poor sleep quality.
Change in Body Mass Index (BMI) | Baseline, End of study (3 months)
  Body mass index (BMI) will be calculated as weight in kilograms divided by height in meters squared from measured height and weight. Measurements of height to the nearest 0.1 cm using A SECA 213 portable stadiometer and weight to the nearest 0.1 kg using a SECA 813 high-capacity weight scale will be conducted in duplicate.
Change in Lipids (non-HDL cholesterol) | Baseline, End of study (3 months)
  Change in lipid levels throughout the study.
Change in HbA1c | Baseline, End of study ( 3 months)
  Change in the HbA1c levels during the study will be reported
Change in Blood pressure | Baseline, Emd of study (3 months)
  Blood pressure (BP) (resting) will be measured three times with a CARESCAPE V100 blood pressure monitor after the participant is seated for five minutes. The average of the last two BP measurements will be used to calculate the mean systolic and diastolic BP.

SECONDARY OUTCOMES:
Social Isolation | Baseline, End of study (3 months)
  Social Isolation will be assessed with the PROMIS Social Isolation SF 8a. Eight items related to perceived feelings of being excluded or disconnected from others are scored on a five-point scale (0-4 = "never" to "always"). Responses are summed to create a raw total score (0-32) that is then rescaled into a standardized score with a mean of 50 and a standard deviation of 10. It has been validated in Latina women
Participant Satisfaction | T1 (1.2 months) ,T2 (3 months), T3 (6 months), T4 (7-9 months)
  Client Satisfaction Questionnaire (CSQ-8), an 8-item scale using a 4-point scale ("quite dissatisfied" to "very satisfied") will be administered to determine the extent to which participants' needs were met
Instrumental support | Baselien, End of study (3 months)
  Instrumental support will be assessed by study documentation of referrals for social needs or SDOH-related factors, CHW resource navigation, and participants' self-report about services offered and services received. We recognize that services offered are not necessarily accepted or received, given participants' autonomy and restraints.
Companionship support | Baseline, End of study (3 months)
  Companionship support will be assessed using the Multidimensional Scale of Perceived Social Support, a 12-item survey to assess three sources of support - Family, Friends, and Romantic Partner
  Each subscale score is the mean of its four items.
  * The total score is the mean of all 12 items.
  * Higher scores indicate greater perceived support.
Informational Support SF 8a | Baseline, End of study (3 months)
  This includes 8 items scored on a five-point scale ("never" to "always")
Emotional Support | Baseline, End of study (3 months)
  This will be assessed using the PROMIS Emotional Support SF 8a, which includes 8 items scored on a five-point scale ("never" to "always").
Gender related stress | Baseline, End of study (3 months)
  Gender-related stress will be assessed with the Hispanic Women's Social Stressor Scale which is a reliable and valid measure of the social stressors experienced by U.S.-born and Mexico-born Hispanic women. It is a 41-item scale with 6 subscales - immigration, socioeconomic, racism-related, familial, parental, and employment
Occupational stress | Baseline, End of study (3 months)
  Occupational stress will be assessed with the Migrant Farmworker Stress Inventory (MFWSI), a 39-item self-report instrument that assesses the quality and severity of stress inherent in migrant farmwork; it was developed for adult migrant farmworkers. The MFWSI requires a 6th-grade literacy level and can be verbally administered if necessary. Each item is scored from 0 to 4. The total MFWSI score is obtained by summing the scores for all 39 items. Possible MFWSI scores range from 0 to 156, with higher scores indicating a greater degree of stress related to the migrant farmworker lifestyle.
Social needs | Baseline. End of study (3 months)
  Social needs/SDOH will be assessed using the Centers for Medicare & Medicaid Services Health-Related Social Needs Tool (HRSN), a 10-item scale covering 5 domains (housing, food, transportation, utilities, and interpersonal safety) with positive responses indicating an associated social need.62 We will assess social needs at baseline and at subsequent timepoints, ask about any changes, and what prompted those changes (participant/CHW initiated or external factor).
Childhood trauma exposure | Baseline, End of study (3 months)
  Childhood trauma exposure will be assessed with the Adverse Childhood Events (ACES) Questionnaire, a 10-item self-report measure of personal experiences of physical, emotional, or sexual abuse or neglect (5 questions) and experiences of adversity related to family members, e.g., mental illness, incarceration, death.25 Each item is scored with one point for each experience. Total scores (number of ACES) are associated with increased risk of toxic stress and health conditions Higher ACE scores correlate with greater risk for chronic diseases, mental health disorders, substance use, and social challenges later in life
Lifetime trauma exposure | Baseline
  Lifetime trauma exposure will be assessed with the Life Events Checklist (LEC-5) -a 17-item measure of lifetime trauma, including type and frequency. Respondents indicate varying levels of exposure to each type of potentially traumatic event included on a 6-point nominal scale, and respondents may endorse multiple levels of exposure to the same trauma type. The LEC-5 does not yield a total score or composite score.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Ferranti, PhD, Principal Investigator — Emory University
Locations (1):
- Southern GA - Colquitt County, Ellenton, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
The shared data will include de-identified quantitative and qualitative data collected through:
  Surveys (social, behavioral, clinical data, including anthropometric and blood pressure measures) Clinical lab results (e.g., lipid panel, Hgb A1c) Transcripts from semi-structured interviews Data analysis files (e.g., SAS, SPSS, R, and MAXQDA outputs) Data dictionaries and supporting metadata
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: De-identified data will be made available no later than the time of publication of primary results or at the end of the funding period, whichever occurs first. Data will remain available indefinitely in the Emory Dataverse for continued public access.
Access Criteria: Data will be shared with qualified investigators who have an appropriate research question and an approved Data Use Agreement (DUA).
  Data may be used for secondary analyses consistent with the original informed consent and within the scope of social, behavioral, and clinical research related to cardiovascular health, social determinants of health, and intervention outcomes.
  Data will be shared through the Emory Dataverse repository. All datasets will be assigned Digital Object Identifiers (DOIs), accompanied by relevant documentation, and made available via secure access mechanisms defined by Emory Dataverse policy